CLINICAL TRIAL: NCT03836690
Title: Phase I Study of Transfer of Effector Memory T Cells (Tem) Following Allogeneic Stem Cell Transplantation
Brief Title: Transfer of Effector Memory T Cells (Tem) Following Allogeneic Stem Cell Transplantation
Acronym: ToTem
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0372; MR/R025436/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2019-01-10; First posted 2019-02-11 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Lymphoma; Leukemia; Myeloma; Myelodysplastic Syndromes; Severe Aplastic Anemia; Primary Immune Deficiency; Graft Vs Host Disease
MeSH Terms: conditions — Lymphoma; Leukemia; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Anemia, Aplastic; Primary Immunodeficiency Diseases; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donor T cells depleted of CD62L+ cells (CD62L- Tem) (Experimental): Donors will undergo a steady state apheresis for the collection of T cells. Selection of CD62L- Tem at the required dose will be performed at UCL Centre for Cell, Gene and Tissue Therapeutics (CCGTT). Donor Tem will be infused into patients on day 24-32 following allo-Stem Cell Transplant.
  Interventions: Biological: CD62L- Tem

INTERVENTIONS:
Biological: CD62L- Tem — Donor memory T cells that have been depleted of CD62L+

SUMMARY:
RATIONALE: Following stem cell transplantation, a major risk is graft-versus-host disease (GVHD). This occurs when donor immune cells that have been infused recognise the host's cells as 'foreign' and attack these cells. Prevention of GVHD relies upon depletion of donor immune T cells or drugs that block T cell function. However, these methods also increase the risk of life threatening infection. There is an important unmet need for better means of accelerating immune recovery following stem cell transplantation while avoiding GVHD.

Pre-clinical studies have shown that infusion of donor CD62L- effector memory T cells (Tem) into the host improve immune recovery after allo-Stem Cell Transplant but do not cause GVHD.

PURPOSE: This phase I dose escalation trial aims to determine the feasibility and safety of transfer of donor Tem following allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Phase I study using a Bayesian Time-to-Event Continual Reassessment Method (CRM) to determine safety and maximum tolerated dose (MTD) of CD62L- Tem.

Eligible patients and HLA-identical sibling donors will be registered prior to stem cell transplant (SCT). Donors will undergo an additional steady state apheresis for the collection of T cells between day -14 and day +24 of the allo-SCT according to logistics. Selection of Tem at the required dose will be performed at UCL Centre for Cell, Gene and Tissue Therapeutics (CCGTT) before distribution of the cryopreserved cells to the trial centre. Doses of Tem selected and infused will be: 1x10^5, 3x10^5, 1x10^6 or 3x10^6.

Donor Tem will be infused on day 24-32 following allo-SCT. Patients will be followed-up for 12 months with specific evaluation points just prior to Tem infusion and at 3, 6, 9 and 12 months following allo-SCT.

ELIGIBILITY:
Patient Registration Inclusion Criteria:

* Severe aplastic anaemia or
* Primary immune deficiency or
* Haematological cancer which can be ONE OF the following:

  * Non-Hodgkin's lymphoma (NHL) in CR or PR;
  * Hodgkin's lymphoma (HL) in CR or PR;
  * Chronic (Pro-)lymphocytic leukaemia (CLL or PLL) in CR or PR
  * Plasma cell myeloma (PCM) in CR, VGPR or PR;
  * Acute myeloid leukaemia (AML) in CR;
  * Acute lymphoblastic leukaemia (ALL) in CR;
  * Myelodysplastic syndrome (MDS) < 10 % blasts in bone marrow;
  * Chronic myelomonocytic leukaemia (CMML) < 10% blasts in bone marrow
* Suitable for HLA-identical sibling transplant using a standard alemtuzumab-based conditioning regimen with calcineurin-inhibitor based immunoprophylaxis
* Aged ≥ 16 years, <70 years
* Written informed consent

Patient Registration Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Life expectancy of < 8 weeks
* Currently taking part in any other interventional clinical research study (involving any IMP, ATMP or cellular therapy)
* Proposed use of any other method of GVHD prophylaxis other than alemtuzumab and calcineurin inhibitor
* Organ dysfunction:

  * LVEF<45%
  * Creatinine >200 µmol/lglomerular filtration rate (corrected) <50ml/min
  * Bilirubin > 50 µmol/l
  * AST or ALT >3x 2.5 x ULN (NB: If both are performed then both must be ≤3 2.5 x ULN)

Patient Trial Treatment Exclusion criteria:

* Prior or active acute pattern GvHD of any grade
* Relapse or progression
* Primary or secondary graft failure
* Has received other cellular therapies

Donor inclusion criteria:

* Aged ≥ 16 years
* HLA-identical sibling
* Have met transplant centre criteria regarding suitability for cell therapy donation
* Negative for HIV 1 and 2, hepatitis B, hepatitis C, HTLV-1 and 2, syphilis serology (to be confirmed before both registration and before trial treatmentat time of or up to 7 days following donation)
* Written informed consent

Donor exclusion criteria:

- Pregnant/lactating women

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity (DLT) | up to 72 days after Tem infusion
  Occurrence of dose limiting toxicity (DLT) (defined as acute-pattern GvHD grade II-IV)

SECONDARY OUTCOMES:
Incidence and severity of acute GvHD | From date of infusion of Tem until 100 days post stem cell transplant
  Incidence and severity of acute GvHD (whether dose limiting or not)
Incidence and severity of chronic GvHD | From date of infusion of Tem up to 1 year post stem cell transplant
  Incidence and severity of chronic GvHD
Non-relapse mortality | From date of patient registration up to 1 year post stem cell transplant
  Death without reoccurrence of cancer
Overall survival | From date of patient registration up to 1 year post stem cell transplant
  Death
Progression-free survival | From date of patient registration up to 1 year post stem cell transplant
  Disease progression or death
Incidence/type of infection requiring inpatient admission | From date of infusion of Tem up to 1 year post stem cell transplant
  Any infection that has required an inpatient admission, incidence and type of infection
Total Number of inpatient days | From date of infusion of Tem up to 1 year post stem cell transplant
  Total Number of inpatient days for any reason

OTHER OUTCOMES:
TCR repertoire analysis by deep CDR3 sequencing | Day -14 to -7 (day of cell processing) and day 100 and 360 post stem cell transplant
Chimerism of immune subsets (analysing the genetic profiles of recipient and donor at baseline and following stem cell transplant) | Pre-Registration and Day 100, 180, 270, 360 post stem cell transplant
  Identifying the genetic profiles of the recipient and of the donor at baseline, evaluating changes in this following stem cell transplant
Assessing the reconstitution level of virus- and bacterial-specific immunity (by measuring the levels of immune cells involved in virus- and bacterial immunity post Tem Infusion) | Day 100, 180, 270, 360 post stem cell transplant
  Measuring the levels of immune cells at specific points in follow up to determine how virus- and bacterial-specific immunity recovers in patients following a stem cell transplant and Tem infusion
Difference between donor immune profile with number of CD62L- Tem selected | Day -14 to -7 (day of cell processing)
  Analysing the donors immune profile pre and post CD62L- Tem selection (cell processing), against the cohort the patient is in (which dose of CD62L- Tem they will receive).
Alemtuzumab levels on the day of CD62L- Tem infusion | Day 28 post stem cell transplant

CONTACTS AND LOCATIONS:
Locations (1):
- UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No